CLINICAL TRIAL: NCT03517566
Title: A Randomized, Double-blind, Placebo-controlled Multicenter Dose Ranging Study to Assess the Safety and Efficacy of Multiple Oral ZPL389 Doses in Patients With Moderate to Severe Atopic Dermatitis (ZEST Trial)
Brief Title: A Study to Assess the Safety and Efficacy of ZPL389 in Patients With Moderate to Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZPL389A2203
Record Dates: First submitted 2018-03-27; First posted 2018-05-07 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; AD; eczema; atopic eczema; itch, pruritus; histamine 4 receptor; antagonist; H4R; ZPL389; ZPL389A2203; dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus; Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- ZPL389 3mg (Experimental): ZPL389 3 mg oral powder
  Interventions: Drug: ZPL389 3mg
- ZPL389 10 mg (Experimental): ZPL389 10 mg oral powder
  Interventions: Drug: ZPL389 10mg
- ZPL389 30mg (Experimental): ZPL389 30 mg oral powder
  Interventions: Drug: ZPL389 30mg
- ZPL389 50mg (Experimental): ZPL389 50 mg oral powder
  Interventions: Drug: ZPL389 50mg

INTERVENTIONS:
Drug: Placebo — once daily from baseline until week 16
  Arms: placebo
Drug: ZPL389 3mg — ZPL389 3 mg oral powder; once daily from baseline to week 16
  Arms: ZPL389 3mg
Drug: ZPL389 10mg — ZPL389 10 mg oral powder; once daily from baseline to week 16
  Arms: ZPL389 10 mg
Drug: ZPL389 30mg — ZPL389 30 mg oral powder; once daily from baseline to week 16
  Arms: ZPL389 30mg
Drug: ZPL389 50mg — ZPL389 50 mg oral powder; once daily from baseline to week 16
  Arms: ZPL389 50mg

SUMMARY:
This was a randomized, double-blind, placebo-controlled, parallel-group study to assess safety and efficacy of ZPL389 in subjects with moderate to severe atopic dermatitis with a total study duration up to 24 weeks

DETAILED DESCRIPTION:
A screening period of up to 4 weeks was followed by a 16-week double blinded treatment period.

After the end of treatment visit, subjects were offered the possibility of ongoing treatment in the extension study (CZPL389A2203E1/ NCT03948334), or of entering the 4 week treatment-free follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give a written, signed and dated informed consent
* Chronic atopic dermatitis present for at least 1 year before Baseline
* Moderate to severe atopic dermatitis defined as per EASI, IGA and BSA.
* Documented recent history (within 6 months before the screening visit) of inadequate response to treatment with topical medications or for whom topical treatments are otherwise medically inadvisable
* Candidate for systemic treatment

Exclusion Criteria:

* Any skin disease that would confound the diagnosis or evaluation of atopic dermatitis disease activity
* Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days or until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
* History of hypersensitivity to any of the study drug constituents or to drugs of similar chemical classes.
* Participation in prior ZPL389 studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (77):
- United States (10):
  - Novartis Investigative Site, Litchfield Park, Arizona
  - Novartis Investigative Site, Fountain Valley, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Fairborn, Ohio
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, West Jordan, Utah
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Leuven, Belgium
- Canada (5):
  - Novartis Investigative Site, Markham, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Sainte-Hyacinthe, Quebec
- Czechia (4):
  - Novartis Investigative Site, Karlovy Vary, Czech Republic
  - Novartis Investigative Site, Nový Jičín, Czech Republic
  - Novartis Investigative Site, Prague, Prague 1
  - Novartis Investigative Site, Prague
- Finland (3):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- Germany (12):
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Osnabrück
- Novartis Investigative Site, Debrecen, Hungary
- Novartis Investigative Site, Kopavogur, Iceland
- Japan (11):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Shinagawa Ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Tokyo
- Netherlands (4):
  - Novartis Investigative Site, Bergen op Zoom
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Rotterdam
- Poland (4):
  - Novartis Investigative Site, Warsaw, Mazowian
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
- Russia (9):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Stavropol
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (4):
  - Novartis Investigative Site, Bardejov, SVK
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Svidník
- Taiwan (2):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Taipei
- United Kingdom (5):
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=723

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 293 subjects randomized at baseline to one of the five treatment arms.
  Two mis-randomized subjects in the placebo arm were excluded from the baseline analysis population.
Period: Overall Study
Arm/Group | Placebo | ZPL389 3mg | ZPL389 10 mg | ZPL389 30mg | ZPL389 50mg
Started | 74 | 37 | 36 | 73 | 73
Completed | 42 | 16 | 21 | 39 | 41
Not Completed | 32 | 21 | 15 | 34 | 32
Not completed — Adverse Event | 5 | 2 | 2 | 8 | 7
Not completed — Lack of Efficacy | 3 | 2 | 1 | 1 | 4
Not completed — Lost to Follow-up | 3 | 1 | 1 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 1 | 0 | 1 | 1
Not completed — Study terminated by Sponsor | 11 | 5 | 6 | 14 | 12
Not completed — Subject Decision /Guardian Decision | 9 | 8 | 5 | 8 | 8

BASELINE CHARACTERISTICS:
Population: All subjects to whom study treatment was assigned. Two Mis-randomized (mis-randomized in Interactive Response Technology (IRT)) subjects in the placebo group were excluded. Mis-randomized subjects were defined as cases where IRT was contacted by the site either prematurely or inappropriately prior to confirmation of the subject's final randomization eligibility and no study medication was administered to the subject.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ZPL389 3mg | ZPL389 10 mg | ZPL389 30mg | ZPL389 50mg | Total
Number analyzed (Participants) | 72 | 37 | 36 | 73 | 73 | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (12.79) | 38.1 (11.86) | 32.1 (9.93) | 34.9 (11.69) | 35.2 (11.91) | 35.0 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 17 | 17 | 32 | 25 | 125
  Male | 38 | 20 | 19 | 41 | 48 | 166
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 51 | 26 | 24 | 55 | 52 | 208
  Black or African American | 0 | 0 | 3 | 3 | 2 | 8
  Asian | 21 | 11 | 9 | 15 | 17 | 73
  Multiple | 0 | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of IGA Responders at Week 16
Description: Investigator's Global Assessment (IGA) score is used to determine the severity of atopic dermatitis symptoms and clinical response to treatment. It reflects a subject's overall disease severity for the whole body. The scale includes 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe. It is a static scale and does not refer to previous status of the subject.
  IGA response is defined as achievement of an IGA score of 0 or 1 with a 2-point reduction from baseline without use of confounding therapy (e.g. rescue medication) up to the assessment time point.
  Treatment discontinuations for lack of efficacy or adverse event are considered non-responders.
  Percentage of responders was calculated based on a logistic regression model with response as outcome variable and treatment (dose as categorical variable) and baseline IGA as covariates.
Time Frame: Week 16
Population: Full analysis set (FAS) comprised all subjects who were randomized and to whom study treatment had been assigned. Mis-randomized subjects (mis-randomized in IRT) were excluded from the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ZPL389 3mg | ZPL389 10 mg | ZPL389 30mg | ZPL389 50mg
Number analyzed (Participants) | 72 | 37 | 36 | 73 | 73
Percentage of participants | 1.9 [-1.6 to 5.3] | 3.3 [-4.3 to 10.9] | 7.2 [-2.3 to 16.8] | 0.8 [-2.0 to 3.7] | 6.9 [0.6 to 13.2]

2. Secondary Outcome: Percent Change From Baseline in EASI Score at Week 16
Description: Eczema Area and Severity Index (EASI) is used to assess the extend and severity of atopic dermatitis on a scale from 0 to 72 where 72 is worst eczema.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | Placebo | ZPL389 3mg | ZPL389 10 mg | ZPL389 30mg | ZPL389 50mg
Number analyzed (Participants) | 72 | 37 | 36 | 73 | 73
Percent change from baseline | -55.0 [-66.9 to -43.1] | -49.4 [-67.4 to -31.4] | -50.7 [-67.3 to -34.1] | -46.2 [-58.8 to -33.6] | -52.7 [-65.0 to -40.4]

3. Secondary Outcome: Percent Change From Baseline in EASI Score Over Time
Description: as for outcome 2
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | Placebo | ZPL389 3mg | ZPL389 10 mg | ZPL389 30mg | ZPL389 50mg
Number analyzed (Participants) | 72 | 37 | 36 | 73 | 73
Percent change from baseline
  Week 2 | -17.1 [-26.6 to -7.5] | -20.1 [-34.2 to -6.1] | -10.3 [-23.8 to 3.1] | -14.2 [-24.0 to -4.3] | -16.7 [-26.4 to -7.1]
  week 4 | -19.7 [-30.6 to -8.9] | -36.1 [-51.4 to -20.9] | -25.6 [-40.6 to -10.7] | -17.7 [-29.0 to -6.4] | -30.0 [-40.6 to -19.4]
  week 6 | -42.8 [-53.0 to -32.6] | -47.6 [-62.3 to -32.9] | -43.2 [-57.3 to -29.0] | -33.2 [-44.0 to -22.3] | -43.5 [-54.0 to -33.0]
  week 8 | -49.3 [-61.1 to -37.4] | -50.1 [-66.8 to -33.4] | -47.4 [-63.9 to -30.9] | -38.1 [-50.5 to -25.7] | -45.5 [-57.4 to -33.6]
  week 12 | -55.4 [-66.0 to -44.8] | -48.7 [-64.2 to -33.2] | -54.1 [-69.2 to -39.1] | -45.1 [-56.4 to -33.8] | -52.7 [-63.7 to -41.7]

4. Secondary Outcome: Percentage of EASI50 Responders Over Time
Description: Eczema Area and Severity Index (EASI) is used to assess the extend and severity of atopic dermatitis on a scale from 0 to 72 where 72 is worst eczema.
  EASI50 response is defined as achieving ≥ 50% improvement (reduction) in EASI score compared to baseline without use of confounding therapy (e.g. rescue medication) up to the assessment time point.
  Treatment discontinuations for lack of efficacy or adverse event are considered non-responders.
  Percentage of responders was calculated based on a logistic regression model with response as outcome variable and treatment (dose as categorical variable) and baseline EASI as covariates
Time Frame: Week 2, Week 4, Week 6, Week 8, Week 12, Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ZPL389 3mg | ZPL389 10 mg | ZPL389 30mg | ZPL389 50mg
Number analyzed (Participants) | 72 | 37 | 36 | 73 | 73
Percentage of participants
  Week 2 | 7.0 [1.1 to 12.9] | 15.0 [3.1 to 27.0] | 12.6 [1.1 to 24.1] | 5.8 [0.3 to 11.2] | 10.1 [3.1 to 17.2]
  week 4 | 13.9 [5.9 to 21.9] | 19.0 [5.4 to 32.5] | 20.1 [6.1 to 34.1] | 9.5 [2.4 to 16.7] | 20.7 [11.4 to 30.1]
  week 6 | 18.4 [9.4 to 27.4] | 15.0 [2.5 to 27.5] | 15.1 [2.5 to 27.7] | 9.5 [2.1 to 16.8] | 16.7 [8.0 to 25.4]
  week 8 | 18.9 [9.7 to 28.0] | 18.0 [4.5 to 31.5] | 16.4 [3.3 to 29.5] | 9.4 [2.2 to 16.6] | 12.8 [4.8 to 20.7]
  week 12 | 20.3 [10.9 to 29.7] | 11.4 [-0.4 to 23.1] | 20.3 [5.8 to 34.9] | 12.6 [4.3 to 20.9] | 12.0 [4.2 to 19.7]
  week 16 | 16.8 [7.9 to 25.8] | 14.4 [1.4 to 27.3] | 22.7 [7.5 to 37.9] | 12.1 [3.9 to 20.3] | 12.7 [4.6 to 20.7]

5. Secondary Outcome: Percentage of EASI75 Responders Over Time
Description: Eczema Area and Severity Index (EASI) is used to assess the extend and severity of atopic dermatitis on a scale from 0 to 72 where 72 is worst eczema.
  EASI75 response is defined as achieving ≥ 75% improvement (reduction) in EASI score compared to baseline without use of confounding therapy (e.g. rescue medication) up to the assessment time point.
  Treatment discontinuations for lack of efficacy or adverse event are considered non-responders.
  Percentage of responders was calculated based on a logistic regression model with response as outcome variable and treatment (dose as categorical variable) and baseline EASI as covariates
Time Frame: Week 2, Week 4, Week 6, Week 8, Week 12, Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ZPL389 3mg | ZPL389 10 mg | ZPL389 30mg | ZPL389 50mg
Number analyzed (Participants) | 72 | 37 | 36 | 73 | 73
Percentage of participants
  week 2 | 0.0 [-0.0 to 0.0] | 0.0 [-3.0 to 4.4] | 0.0 [-3.1 to 4.4] | 1.4 [-1.3 to 4.1] | 1.5 [-1.4 to 4.3]
  week 4 | 2.8 [-1.0 to 6.6] | 7.0 [-2.0 to 16.0] | 1.7 [-3.9 to 7.2] | 1.8 [-1.6 to 5.2] | 1.4 [-1.3 to 4.2]
  week 6 | 5.6 [0.3 to 10.9] | 10.3 [-0.4 to 21.0] | 7.1 [-1.9 to 16.1] | 1.8 [-2.0 to 5.7] | 7.4 [1.2 to 13.6]
  week 8 | 6.0 [0.4 to 11.6] | 10.9 [-0.2 to 21.9] | 8.5 [-1.8 to 18.8] | 2.5 [-1.8 to 6.8] | 6.1 [0.4 to 11.9]
  week 12 | 4.6 [-0.4 to 9.6] | 6.2 [-3.1 to 15.6] | 10.6 [-0.9 to 22.0] | 2.8 [-1.6 to 7.2] | 5.8 [-0.0 to 11.7]
  week 16 | 9.7 [2.6 to 16.8] | 7.1 [-2.8 to 16.9] | 12.9 [0.3 to 25.5] | 3.1 [-1.7 to 7.8] | 9.3 [2.1 to 16.6]

6. Secondary Outcome: Percentage of IGA Responders Over Time
Description: as for outcome 1
Time Frame: Week 2, Week 4, Week 6, Week 8, Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | ZPL389 3mg | ZPL389 10 mg | ZPL389 30mg | ZPL389 50mg
Number analyzed (Participants) | 72 | 37 | 36 | 73 | 73
Percentage of participants
  week 2 | 0.0 [-0.0 to 0.0] | 2.7 [-2.5 to 7.9] | 0.0 [-0.7 to 0.8] | 0.0 [-0.0 to 0.0] | 0.0 [-0.0 to 0.0]
  week 4 | 0.0 [-0.0 to 0.0] | 2.8 [-2.6 to 8.3] | 0.0 [-1.4 to 1.6] | 0.0 [-0.6 to 0.7] | 0.0 [-0.4 to 0.4]
  week 6 | 1.4 [-1.3 to 4.1] | 6.1 [-2.1 to 14.4] | 5.9 [-2.0 to 13.8] | 0.0 [-1.9 to 2.9] | 0.0 [-1.2 to 1.6]
  week 8 | 1.6 [-1.4 to 4.5] | 3.8 [-3.1 to 10.7] | 6.5 [-2.1 to 15.0] | 0.0 [-1.7 to 2.7] | 2.0 [-1.6 to 5.6]
  week 12 | 1.5 [-1.4 to 4.4] | 4.0 [-3.3 to 11.3] | 5.6 [-3.1 to 14.2] | 1.9 [-1.6 to 5.5] | 1.0 [-2.1 to 4.1]

7. Secondary Outcome: Number of Patients With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject after providing written informed consent for participation in the study until the end of study visit. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
Time Frame: Up to week 20
Population: Safety Set included all subjects who received at least one dose of study medication. Subjects were analyzed according to treatment received. The safety analyses were based on safety sets (SAF).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ZPL389 3mg | ZPL389 10 mg | ZPL389 30mg | ZPL389 50mg
Number analyzed (Participants) | 72 | 37 | 36 | 73 | 73
Participants
  AE | 44 | 22 | 18 | 48 | 43
  SAE | 2 | 1 | 3 | 1 | 3
  AEs leading to discontinuation | 7 | 3 | 2 | 11 | 12

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 4 weeks post treatment, up to maximum duration of 20 weeks
Description: Any sign or symptom that occurs during the study treatment plus the 4 weeks post treatment
Groups:
- ZPL389 3 mg: ZPL389 3 mg oral powder
- ZPL389 30 mg: ZPL389 30 mg oral powder
- ZPL389 50 mg: ZPL389 50 mg oral powder
- All Patients: All Patients
Arm/Group | Placebo | ZPL389 3 mg | ZPL389 10 mg | ZPL389 30 mg | ZPL389 50 mg | All Patients
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/37 | 0/36 | 0/73 | 0/73 | 0/291
Serious Adverse Events (participants affected / at risk) | 2/72 | 1/37 | 3/36 | 1/73 | 3/73 | 10/291
Other Adverse Events (participants affected / at risk) | 27/72 | 14/37 | 8/36 | 30/73 | 26/73 | 105/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | ZPL389 3 mg (N=37) | ZPL389 10 mg (N=36) | ZPL389 30 mg (N=73) | ZPL389 50 mg (N=73) | All Patients (N=291)
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Herpes dermatitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Risk of future pregnancy miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 1 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | ZPL389 3 mg (N=37) | ZPL389 10 mg (N=36) | ZPL389 30 mg (N=73) | ZPL389 50 mg (N=73) | All Patients (N=291)
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 5 | 9
Influenza like illness (General disorders) | 1 | 0 | 2 | 3 | 3 | 9
Nasopharyngitis (Infections and infestations) | 8 | 2 | 2 | 4 | 4 | 20
Rhinitis (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2 | 6 | 1 | 12
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1 | 3 | 6
Headache (Nervous system disorders) | 5 | 1 | 1 | 2 | 4 | 13
Insomnia (Psychiatric disorders) | 0 | 2 | 1 | 1 | 1 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 3 | 1 | 8
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 11 | 6 | 2 | 14 | 8 | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-09-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT03517566/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT03517566/SAP_002.pdf